CLINICAL TRIAL: NCT06619522
Title: A Phase 2 Study of INCB57643 (BET Inhibitor) in Combination With Ruxolitinib in JAK Inhibitor-naïve Patients With Myelofibrosis
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: 0 participant accrual
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-1031; NCI-2024-08192 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2024-09-25; First posted 2024-10-01 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Myelofibrosis
MeSH Terms: conditions — Primary Myelofibrosis | interventions — ruxolitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- INCB+ R (Experimental)
  Interventions: Drug: Ruxolitinib; Drug: INCB57643

INTERVENTIONS:
Drug: Ruxolitinib — Given orally
Drug: INCB57643 — Given orally

SUMMARY:
To assess INCB05643 + ruxolitinib JAKi-naive patients with myelofibrosis

DETAILED DESCRIPTION:
Primary Objective:

To evaluate splenic response rate by imaging after 24 weeks of treatment.

Secondary Objectives:

To evaluate splenic response rate by imaging after 24 weeks of treatment. To evaluate splenic response rate by imaging after 12 weeks of treatment To evaluate splenic response rate by imaging after 12 weeks of treatment To evaluate the overall splenic response rate and the duration of splenic response To evaluate the overall splenic response rate and the duration of splenic response To evaluate the proportion of patients who achieve both a splenic response and a ≥ 50% reduction in TSS after 24 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Adult (aged ≥ 18 years). Because no dosing or adverse event data are currently available on the use of ruxolitinib in combination with INC057643 in patients <18 years of age, children are excluded from this study.
2. Patients with confirmed diagnosis of MF who meet all of the following criteria:

   1. DIPSS-plus (see Appendix 3) risk category of intermediate-1, intermediate-2, or high
   2. Platelet count ≥100 × 109/L without the assistance of thrombopoietic factors or transfusions
   3. ANC ≥1 × 109/L without the assistance of granulocyte growth factors
   4. Spleen volume of ≥450 cm3 by MRI/CT or spleen length ≥5 cm below the left costal margin
   5. Peripheral blood blast count <10% at the screening hematology assessment
   6. At least 2 symptoms that are measurable (each with a score 3) or 1 symptom with a score of 5 or a total symptom score of 10 using the MFSAF v4.0
   7. No prior treatment with JAKi or BETi allowed
3. ECOG performance status ≤ 2 (Appendix 1)
4. Life expectancy of >24 weeks
5. Serum total bilirubin ≤1.5 × ULN (total bilirubin >1.5 × ULN is acceptable if direct bilirubin ≤ 1.2 × ULN or with a diagnosis of Gilbert's syndrome)
6. AST and ALT ≤2.5 × ULN. The AST and /or ALT may be elevated up to 5 × ULN if the elevation can be reasonably ascribed to liver involvement.
7. Calculated or measured CrCl ≥50 mL/min (either measured or estimated by the Cockcroft- Gault formula) {Cockcroft-Gault formula for eCrCl: eCrCl = (140 - Age) × Mass (kg) × [0.85 if Female]/ 72 × Serum Creatinine (mg/dL)} or GFR ≥50 ml/min/1.73 m2 calculated by the Modification of Diet in Renal Disease formula.
8. Patients must have fully recovered from major surgery and from the acute toxic effects of prior chemotherapy and radiotherapy (residual CTCAE Grade 1 toxicity, e.g., Grade 1 peripheral neuropathy, and residual alopecia are allowed).
9. Both male and female patients and partners of patients, with reproductive potential, must agree to use at least one highly effective contraceptive method while on study therapy and for 90 days after the last dose of INCB057643 for male patients and male partners of female patients, and for 180 days after the last dose of study drug for female patients and female partners of male patients. NOTE: Patients may consider seeking information from the study investigator regarding donation and cryopreservation of germ cells prior to treatment. Male patients should be informed of the risk of testicular toxicity and provided with adequate advice regarding sperm preservation.
10. Patients must give written informed consent to participate in this study before the performance of any study-related procedure.

Exclusion Criteria:

1. Prior treatment with a BET inhibitor.
2. Prior treatment with a JAK inhibitor, including ruxolitinib.
3. Patients who have had a prior splenectomy.
4. Patients who have had splenic irradiation within 6 months of starting study treatment.
5. Current known active or chronic infection with TB, HIV, Hepatitis B, or Hepatitis C. Screening of patients with serologic testing for these viruses is not required. However, patients who have a past history of viral hepatitis or in whom there is a current suspicion of viral hepatitis should have DNA/RNA testing for Hepatitis B and Hepatitis C performed to determine whether there is any current evidence for ongoing infection with these viruses. Patients considered to be at risk for HIV infection should have HIV testing performed. Testing for COVID-19 is not mandatory during the screening for this study. However, based on the local epidemiologic situation and each patient's individual COVID-19 exposure risk and/or vaccination status, investigators should consider testing and in the case of COVID-19 positivity consider delaying the start of the study treatment until the infection is resolved.
6. Patients with active clinically significant infection will not be eligible for enrollment until recovery for at least 2 weeks prior to the first dose of study drug.
7. Patients with anemia deemed clinically significant by the investigator from iron deficiency, B12 and folate deficiencies, or hemolytic anemia.
8. Patient with a major bleeding event causing a decrease in Hgb of ≥2g/dL or leading to transfusion of ≥2 units of packed red cells in the last 6 months prior to enrollment.
9. Patients with liver cirrhosis Child-Pugh Class B or C (see Appendix 4).
10. Patients with rare hereditary problems of galactose intolerance, the Lapp lactase deficiency, or glucose-galactose malabsorption or patients with hypersensitivity to any ingredient in the formulation of ruxolitinib.
11. Patients who have or have had progressive multifocal leukoencephalopathy (PML).
12. Ongoing uncontrolled hypertension despite maximal antihypertensive treatment.
13. Any other concurrent severe and/or uncontrolled concomitant medical condition that in the opinion of the investigator could compromise participation in the study or analysis of study data. This includes but is not limited to clinically significant pulmonary disease or neurological disorders, or active or uncontrolled infections.
14. Systemic anticancer treatment other than hydroxyurea (HU) and anagrelide (ANA) less than 2 weeks (or 5 half-lives, whichever is longer) before the first dose of study treatment. NOTE: HU and ANA are permitted to be used up to 72 hours prior to start of study drugs.
15. Any investigational agent (whether for cancer treatment or not) less than 2 weeks (or 5 half-lives, whichever is longer) before the first dose of study treatment. < 6 weeks for mitomycin-C or nitrosourea.
16. Hematopoietic growth factor (granulocyte growth factor, erythropoiesis stimulating agent, thrombopoietin mimetic) or androgenic steroids less than 4 weeks before the first dose of study drug.
17. Participants with laboratory values at screening defined in Table 18.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-09-11 (Actual); Primary Completion 2025-05-09 (Actual); Study Completion 2025-05-09 (Actual)

PRIMARY OUTCOMES:
Safety and Adverse Events (AEs). Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability]) | Through study completion; an average of 1 year
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Mahesh Swaminathan, MBBS, Principal Investigator — M.D. Anderson Cancer Center

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org